CLINICAL TRIAL: NCT00691145
Title: A Long-term, Non-comparative, Multi-centre Study to Evaluate the Efficacy and Safety of 0.1% and 0.03% Tacrolimus (FK506) Ointment Administered in Adults With Moderate to Severe Atopic Dermatitis FG-506-06-IT-01
Brief Title: Study to Evaluate the Efficacy and Safety of 0.1% and 0.03% Tacrolimus Ointment Administered in Adults With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-06-IT-01
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic dermatitis; Tacrolimus ointment
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment

INTERVENTIONS:
Drug: tacrolimus ointment — transdermal
  Other Names: FK506 ointment

SUMMARY:
The objective of this study is to assess the efficacy and safety of 0.1% and 0.03% Tacrolimus ointment for 12 months in adults with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
The main phase is 6 months duration, but the follow up phase up to 12 months will allow the collection of efficacy and safety data in a period which will include all seasons in each patient, to account for seasonal variability which strongly affect atopic dermatitis course.

ELIGIBILITY:
Inclusion Criteria:

* Patient may be male or female of any ethnic group
* Patient without restricted legal competence, and suffers from moderate to severe atopic dermatitis (Rajka/Langeland score of at least 4.5)
* Patient known to be responsive to topical steroids
* Patient is capable of understanding the purposes and risks of the trial and has given written Informed Consent
* Female patients of childbearing potential must agree to maintain adequate birth control practice during the trial period and during the first four weeks after the end of the study
* Patient meets the following criteria:

  * Topical corticosteroids
  * Systemic corticosteroids (for the treatment of AD only)
  * Systemic non-steroidal immunosuppressants (e.g. cyclosporine, methotrexate)
  * Other investigational drugs
  * Light Treatments (UVA, UVB)
* Patient has not taken and agrees not to take for the complete study period any medication or therapy prohibited by the protocol

Exclusion Criteria:

* Patient has a genetic epidermal barrier defect such as Netherton's syndrome or generalised erythroderma
* Patient is pregnant or breast-feeding
* Patient has a skin infection on the affected (and to be treated) area
* Patient has a known hypersensitivity to macrolides in general, to tacrolimus or any excipient of the ointment
* Patient is simultaneously participating in any other drug trial or less than 28 days have passed between the end of the previous trial and this one
* Any form of substance abuse (including drug or alcohol abuse),psychiatric disorder or condition which, in the opinion of the investigator, may invalidate the communication with the investigator
* Patient is known to be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2002-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The rate of patients with at least 50% (i.e. at least moderate) improvement according to the physician's global evaluation of clinical response at month 6/end of study (if before month 6) visit | 1 year

SECONDARY OUTCOMES:
The rate of patients with at least 50%(i.e. at least moderate) improvement according to the physician's global evaluation of clinical response at month 12/end of study (if after month 6) visit | 1 year
The rate of patients with at least 60% improvement in the Score In Atopic Dermatitis (SCORAD) at month 6/end of study visit (if before month 6) and at month 12/end of study (if after month 6) visit, each compared to baseline (day 1) | 1 year
The incidence of adverse events during the study, including all clinically significant laboratory values | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (25):
- Italy (25):
  - S. Giovanni Rotondo, Foggia
  - Battipaglia, Salerno
  - Ancona
  - Bari
  - Benevento
  - Bergamo
  - Bolzano
  - Catania
  - Genova
  - Mantova
  - Merano
  - Messina
  - Milan
  - Napoli
  - Novara
  - Parma
  - Pavia
  - Perugia
  - Reggio Emilia
  - Roma
  - Sassari
  - Siena
  - Torino
  - Trieste
  - Venezia